CLINICAL TRIAL: NCT00842686
Title: Preoperative Radiotherapy With Capecitabine and Bevacizumab in Locally Advanced Rectal Cancer: CRAB Phase II Study
Acronym: CRAB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Velenik Vaneja, MD, PhD, Institute of Oncolg Ljubljana, Slovenia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21901
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: rectal cancer; capecitabine; bevacizumab; radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab, capecitabine — bevacizumab 5mg/kg days -15,1,15,29 capecitabine 1250 mg/square m/day during radiotherapy radiotherapy 50,4 Gy (1,8 Gy per fraction)
  Other Names: Avastin; Xeloda; radiation

SUMMARY:
The use of preoperative chemoradiation and adjuvant chemotherapy with 5-FU based chemotherapy reduced local recurrence rate to less than 10%, but has only had limited effect on overall survival due to the constantly high (more than 30%) rate of distant metastasis.

However, it has been shown that complete eradication of the primary tumour observed in the histopathological specimen (pathological complete response, pCR) correlates with a favourable overall prognosis so obtaining a pCR might be beneficial. The aim of the study is to investigate whether the addition of bevacizumab to preoperative fluoropyrimidinebased chemoradiation improves pathological complete remission rate in locally advanced rectal cancer with acceptable toxicity. Secondary objectives are to evaluate pathological downstaging rate, histopathological R0 resection rate,sphincter preservation rate, perioperative surgical complication rate, local control, DFS, OS, late toxicity and quality of life.

DETAILED DESCRIPTION:
* radiotherapy: 45 Gy to the pelvis (25x 1.8 Gy on days 1-33, excluding weekends) plus 5.4 Gy on days 36-38 as a boost to the primary tumour (3 fractions of 1.8 Gy).Three- dimensional CT planing and a four field box technique with high energy photons (15 MV) will be used. All fields will be treated daily. Multileaf collimators will be used to shape individual radiation fields. Patients will be irradiated in a prone position with a full bladder and by using belly board to minimize exposure of the small bowel.
* capecitabine 825 mg/m² p.o. twice daily on days 1-38 (including weekends),
* bevacizumab: at dose 5 mg/kg on days -14, 2, 16,30.
* Radical surgery (TME): to be undertaken ideally 6-8 weeks following completion of chemoradiation.

Postoperative treatment (in patients achieving histopathological R0 or R1 resection):capecitabine 1250 mg/m² p.o. twice daily for 14 consecutive days every three weeks; 4 cycles (R0)or 6 cycles (R1) beginning 6-8 weeks after surgery

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with histologically proven adenocarcinoma of the rectum (tumour located below the peritoneum), T3/4 or any node positive disease (clinical stage according the TNM classification system)
* No evidence of metastatic disease.
* The disease must be considered either resectable at the time of entry or thought to become resectable after preoperative chemoradiation.
* Age 18 - 80 years
* WHO Performance Status 0-2
* No prior radiotherapy, chemotherapy or any targeting therapy for rectal cancer
* Adequate hematological, hepatic and renal function Ability to swallow tablets
* Signed informed consent
* Patients must be willing and able to comply with the protocol for duration of the study

Exclusion Criteria:

* Malignancy of the rectum other than adenocarcinoma
* Any unrested synchronous colon cancer
* Other co-existing malignancy or malignancy within the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
* Significant heart disease (uncontrolled hypertension despite of medication (> 150/100 mmHg), NYHA class III or IV heart disease,unstable angina or myocardial infarction within the past 1 year prior the study entry, history of significant ventricular arrhythmia requiring treatment)
* Serious, non-healing wound, ulcer or bone fracture
* Evidence of active peptic ulcer or upper GI bleeding
* Evidence of bleeding diathesis or coagulopathy
* Chronic daily treatment with high-dose aspirin(>325mg/day)
* Current or recent (>10 days) use of full-dose of parenteral anticoagulants or thrombolytic agents for therapeutic purpose
* Patients receiving a concomitant treatment with drugs interacting with capecitabine such as flucitosine, phenytoin, or warfarin
* Known dihydropyrimidine dehydrogenase (DPD)deficiency
* Major surgery within 4 weeks prior to study treatment starts, or lack of complete recovery from the effects of major surgery or open biopsy
* Known hypersensitivity to biological drugs
* Treatment with any investigational drug within 30 days before beginning treatment with the study drug
* Pregnant or lactating patient
* Females with a positive or no pregnancy test unless childbearing potential can be otherwise excluded (amenorrheic for at least 2 years,hysterectomy or oophorectomy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | after pathological examination of surgical speciments

SECONDARY OUTCOMES:
Pathological response rate | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Rate of sphincter sparing surgical procedure | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Histopathological R0 resection rate | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Acute and late toxicity | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Loco-regional failure rate | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Disease-free survival | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Overall survival | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
Quality of life | Toxicity/safety:during preoperative treatment, early and late postoperative follow up

CONTACTS AND LOCATIONS:
Overall Officials: Vaneja Velenik, MD, PhD, Principal Investigator — Institute of Oncology, Ljubljana, Slovenia
Locations (1):
- Onstitute of Oncology, Zaloška 2, Ljubljana, Slovenia

REFERENCES:
- [Background] Camma C, Giunta M, Fiorica F, Pagliaro L, Craxi A, Cottone M. Preoperative radiotherapy for resectable rectal cancer: A meta-analysis. JAMA. 2000 Aug 23-30;284(8):1008-15. doi: 10.1001/jama.284.8.1008. PMID 10944647
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Velenik V, Anderluh F, Oblak I, Strojan P, Zakotnik B. Capecitabine as a radiosensitizing agent in neoadjuvant treatment of locally advanced resectable rectal cancer: prospective phase II trial. Croat Med J. 2006 Oct;47(5):693-700. PMID 17042060
- [Background] Duda DG, Jain RK, Willett CG. Antiangiogenics: the potential role of integrating this novel treatment modality with chemoradiation for solid cancers. J Clin Oncol. 2007 Sep 10;25(26):4033-42. doi: 10.1200/JCO.2007.11.3985. PMID 17827451
- [Background] Willett CG, Boucher Y, Duda DG, di Tomaso E, Munn LL, Tong RT, Kozin SV, Petit L, Jain RK, Chung DC, Sahani DV, Kalva SP, Cohen KS, Scadden DT, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Shellito PC, Mino-Kenudson M, Lauwers GY. Surrogate markers for antiangiogenic therapy and dose-limiting toxicities for bevacizumab with radiation and chemotherapy: continued experience of a phase I trial in rectal cancer patients. J Clin Oncol. 2005 Nov 1;23(31):8136-9. doi: 10.1200/JCO.2005.02.5635. No abstract available. PMID 16258121
- [Background] Czito BG, Bendell JC, Willett CG, Morse MA, Blobe GC, Tyler DS, Thomas J, Ludwig KA, Mantyh CR, Ashton J, Yu D, Hurwitz HI. Bevacizumab, oxaliplatin, and capecitabine with radiation therapy in rectal cancer: Phase I trial results. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):472-8. doi: 10.1016/j.ijrobp.2007.02.001. PMID 17498568